CLINICAL TRIAL: NCT04762940
Title: EFFECTIVENESS OF INTENSIVE TREATMENT WITH ROBOTIC PLUS VIBRATION TO SENSITIVITY AND FUNCTIONALITY REHABILITATION IN STROKE PATIENTS
Brief Title: INTENSIVE TREATMENT WITH ROBOTIC PLUS VIBRATION IN STROKE
Acronym: VIBRAROBOT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Josue Fernandez Carnero, Clinical Professor, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: URJC-MADROÑOS
Record Dates: First submitted 2021-02-12; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Stroke; Activities, Motor; Quality of Life; Sensitivity; Upper Extremity Paresis
Keywords: Stroke; Rehabilitation; Upper limb; Sensitivity; Motor rehabilitation
MeSH Terms: conditions — Stroke; Motor Activity; Hypersensitivity; Paresis

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Assessments will be made by researches blinded for the patient´s group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): They will receive 24 robotics sessions with Amadeo robot three times a week for movement, but without specifically receiving vibration therapy.
  Interventions: Device: Robotic
- Experimental group (Experimental): They will recieve three times a week with 24 sessions plus vibration duration of approximately 20 minutes with a high vibration frequency. Vibration therapy, with proprioceptive stimuli through sensors placed on the distal phalanges of the fingers, modulation from lower to higher frequency being possible will be conducted prior to robotic treatments with Amadeo.
  Interventions: Device: Robotic; Device: Vibration

INTERVENTIONS:
Device: Robotic — The Amadeo® Manual Robotic System (Tyromotion GmbH, Graz, Austria) is designed for rehabilitative treatment of the hand and fingers providing robot-assisted exercise for the finger flexors and extensors. This system has a controlled position, active, active-assisted and passive exercise mode, it also allows isometric exercises with visual feedback provided during computerized games that emphasize flexion and extension.
  Robotic treatment will be conducted three times a week with 24 sessions (a month and a half of treatment) with assisted therapy: It allows to carry out the movement by force of the fingers themselves, compensating the range of movement that the user does not perform; and interactive therapy: it allows to carry out active finger movement oriented to tasks or games. These can be configured to adapt them as much as possible to the capabilities of the user.
Device: Vibration — Vibration duration of approximately 20 minutes with a high vibration frequency will be conducted prior to robotic treatment. The intensity and timing of this treatment has been based on previous protocols, as previously justified in this project. Vibration therapy, with proprioceptive stimuli through sensors placed on the distal phalanges of the fingers, modulation from lower to higher frequency being possible (high frequency vibration of 300 Hz).
  Arms: Experimental group

SUMMARY:
The Amadeo® Manual Robotic System (Tyromotion GmbH, Graz, Austria) is designed for rehabilitative treatment of the hand and fingers providing robot-assisted exercise for the finger flexors and extensors. This system has a controlled position, active, active-assisted and passive exercise mode, it also allows isometric exercises with visual feedback provided during computerized games that emphasize flexion and extension. Another of the functions that this device presents and that differentiates it from other handheld robotic systems is its vibration function. Through sensors that are placed on the fingertips, providing a vibratory proprioceptive stimulus of different frequencies.

Currently, there are no published trials on the efficacy of the vibration of this device and its consequent improvement in the sensitivity and functionality of patients with hemiparesis after stroke. Investigations have been conducted in patients with peripheral lesions and in the healthy population. A preliminary study with monkeys demonstrated that the frequency of the vibration presents better results when the muscle stretch receptors are driven by a high frequency vibration, activating the neurons corresponding to the motor cortex and in the 3rd primary sensory area. More recent studies have shown the efficacy of focal vibratory stimulation applied to the wrist and forearm muscles, specifically the application to the tendon of the stimulated muscle.

Regarding the most appropriate form of stimulation, the most important determining factors to highlight are the frequency of application, the duration and intensity and the time of application. The mechanism of action of local muscle vibration is to stimulate various receptors. Meissner corpuscles respond best around 40 Hz, while Vater-Pacini corpuscles around 100 Hz. Together, they are also known as rapidly adapting cutaneous receptors. In contrast, Merkel-Ranvier cells and Ruffini corpuscles are called slow-adapting and classically described as sensitive to sustained pressure. That is why authors of different studies have focused on high frequency vibration of 300 Hz, for 30 minutes. 3 times per week. The duration of vibratory stimulation, different studies show the effects of vibration and changes in the cortex after performing the treatment constantly, for about ten days, intensively three to four days a week, observing long-term changes in terms on cortical excitability.

DETAILED DESCRIPTION:
The rehabilitation of the stroke patient is an individual process, adapted to each type of patient, continuous and oriented by objectives whose main purpose is to treat and / or compensate for deficits and disability to achieve the maximum functional independence achievable in each case, facilitating independence and reintegration into the family, social and work environment. The stroke rehabilitation program is a complex process that requires a multidisciplinary approach to existing motor, sensory and / or neuropsychological deficiencies through re-education techniques based fundamentally on the phenomenon of neuronal plasticity and task-oriented rehabilitation.

There is evidence that supports the need to work on the intensity and repetition of motor skills in treatments to promote neuroplasticity and motor relearning. Considering the significant advances in information and communication technology (ICT) and more specifically the rapid development and deployment of technology, a number of recent systematic and non-systematic reviews highlight the increasing use of wearable devices to provide intensity to rehabilitation after of suffering a stroke including robotics, virtual reality, functional electrical stimulation (FES).

Robot-assisted therapy for post-stroke rehabilitation is relatively new as a complementary tool to physical therapy, through which patients practice their limb and paretic hand, resorting to or resisting the force offered by these robots.

The strongest point of these devices is the "attractive" variety of exercises that provide the user with great motivation, in addition to the "intensity" factor in the therapies. These factors allow for rehabilitation treatments with robotic technology, which cannot be achieved with any conventional rehabilitation therapy. The Amadeo® Manual Robotic System (Tyromotion GmbH, Graz, Austria) is designed for rehabilitative treatment of the hand and fingers providing robot-assisted exercise for the finger flexors and extensors. This system has a controlled position, active, active-assisted and passive exercise mode, it also allows isometric exercises with visual feedback provided during computerized games that emphasize flexion and extension.

Another of the functions that this device presents and that differentiates it from other handheld robotic systems is its vibration function. Through sensors that are placed on the fingertips, providing a vibratory proprioceptive stimulus of different frequencies.

Currently, there are no published trials on the efficacy of the vibration of this device and its consequent improvement in the sensitivity and functionality of patients with hemiparesis after stroke. Investigations have been conducted in patients with peripheral lesions and in the healthy population. A preliminary study with monkeys demonstrated that the frequency of the vibration presents better results when the muscle stretch receptors are driven by a high frequency vibration, activating the neurons corresponding to the motor cortex and in the 3rd primary sensory area. More recent studies have shown the efficacy of focal vibratory stimulation applied to the wrist and forearm muscles, specifically the application to the tendon of the stimulated muscle.

Regarding the most appropriate form of stimulation, the most important determining factors to highlight are the frequency of application, the duration and intensity and the time of application. The mechanism of action of local muscle vibration is to stimulate various receptors. Meissner corpuscles respond best around 40 Hz, while Vater-Pacini corpuscles around 100 Hz. Together, they are also known as rapidly adapting cutaneous receptors. In contrast, Merkel-Ranvier cells and Ruffini corpuscles are called slow-adapting and classically described as sensitive to sustained pressure. That is why authors of different studies have focused on high frequency vibration of 300 Hz, for 30 minutes. 3 times per week.

The duration of vibratory stimulation, different studies show the effects of vibration and changes in the cortex after performing the treatment constantly, for about ten days, intensively three to four days a week, observing long-term changes. term on cortical excitability. With regard to the evaluation of the different variables that are the subject of this study, a review of the tests has been carried out with more sensitive and reliable results at present. The Fugl Meyer Assessment Upper Extremity Scale (UE) continues to be one of the most commonly used and specific tests to assess motor and sensory impairment in stroke patient.

Since one of the main variables and object of measurement of the present study is sensitivity, it has been introduced, Semmes-Weinstein® Monofilaments is the most common and accurate instrument for sensory assessment. There are multiple scales to measure functionality such as FIM36 (Functional Independence Measure), FAM (Functional Assessment Measure), Barthel Index, however, the Motor Activity Log scale measures the functionality and motor performance of the most affected upper limb in a specific way, as well as its spontaneous use and integration in quantity and quality in the performance of Activities of Daily Living.

Stroke impact Scale (SIS) is a specific questionnaire for patients with brain damage and measures the impact it has had on their quality of life. SIS version 3.0 contains 8 domains related to hand function, strength, activities of daily living, communication, emotion, memory, and thinking. The SIS is a valid and reliable measure for a diverse group of patients after suffering a stroke.

The present study aims to determine, in stroke patients with left hemiparesis, the efficacy of intensive vibration therapy treatment with the Amadeo® robotic system, focusing on assessing sensitivity, integration of the affected upper limb and functionality, as well such as the improvement in the quality of life in the execution of their Activities of daily living in comparison with those patients who do not receive intensive vibration treatment but do perform upper limb treatment with the Amadeo® robotic system.

We present a randomized controlled trial to compare the improvement in sensitivity, the integration of the hemibody and the functionality in a sample of people who have suffered a stroke with left hemiparesis and receive intensive vibratory treatment, through the Amadeo robotic system ® compared to another population with the same characteristics that does not receive this vibration therapy, although they do perform robotic treatment without vibration.

It will be conducted at the "Los Madroños" hospital and Clínica NEURON (Madrid, Spain).

Inclusion criteria:

* Age: people aged between 30 and 80 years.
* Diagnosis: stroke in the right hemisphere.
* Right-handed.
* Present hemiparesis or left hemiplegia with paralysis / paresis in his affected hand.
* People with sensitivity alterations as a result of stroke.
* Evolution: subacute patients (from three months to one year, and who at the same time meet the subacute criteria of the IMSERSO document of the model of care for people with brain damage, as well as chronic patients (after one year, and who meet the chronicity criteria of the IMSERSO document of the model of care for people with brain damage).
* People without other concomitant pathologies that affect mobility and / or sensitivity
* The acceptance and signing of the informed consent by the user.
* Present a score equal to or greater than 24 points in the Mini-Mntal State Examination (MMSE).
* Patients can be admitted or outpatient as long as they meet the above criteria and belong to the advanced neurorehabilitation unit.

Exclusion criteria:

* Patients with Aphasia and / or Apraxia.
* Patients with serious difficulties in communication.
* Patients who do not present limitation of mobility and / or sensitivity.
* Other concomitant diseases.
* Diagnosis: left or posterior hemisphere stroke.
* Present a score of less than 24 points on the MMSE.
* Age over 80 years and under 30 years.
* The non-acceptance and signing of the informed consent by the subject.
* Evolution: acute patients less than three months of evolution.

Patients eligible to receive treatment will be consecutively randomized into two groups, those who receive robotic therapy with vibration and movement, and those who receive only vibration.

Outcomes:

* Clinical information: patient's sociodemographic data and anamnesis, the neurological examination and the different functional and sensitivity scales of which are:
* Semmes-Weinstein (SW) ® monofilaments for sensitivity assessment
* Fugl Meyer Assessment scale for the upper limb.
* Motor Activity Log (MAL).
* Stroke Impacte Scale (SIS).
* Questionnaire of satisfaction with technology. (based on the principles of the Likert scale)

Follow up:

One month after the post-treatment evaluation, the research team will re-evaluate, administering all the tests from the previous evaluations except for the technology satisfaction questionnaire. It will be carried out in the Advanced Neurorehabilitation Unit and exclusively to the population of the experimental group to see if the results obtained in the treatment are maintained over time.

Intervention:

The patients will be referred by the team made up of rehabilitation doctors and specialized neurologists from Hospital Los Madroños and Clínica NEURON and will receive treatment in its Advanced Neurorehabilitation Units:

* In the "experimental" group, sessions will be held three times a week with 24 sessions (a month and a half of treatment), with a vibration duration of approximately 20 minutes with a high vibration frequency. The intensity and timing of this treatment has been based on previous protocols, as previously justified in this project. Vibration therapy, with proprioceptive stimuli through sensors placed on the distal phalanges of the fingers, modulation from lower to higher frequency being possible
* In the "control" group, they will receive the same 24 robotics sessions three times a week for movement, but without specifically receiving vibration therapy. Therapy will be based on movements.
* Robotic treatment:

Assisted therapy: It allows to carry out the movement by force of the fingers themselves, compensating the range of movement that the user does not perform.

Interactive therapy: Allows to carry out active finger movement oriented to tasks or games. These can be configured to adapt them as much as possible to the capabilities of the user.

ELIGIBILITY:
Inclusion Criteria:

* Age: people aged between 30 and 80 years.
* Diagnosis: stroke in the right hemisphere.
* Right-handed.
* Present hemiparesis or left hemiplegia with paralysis / paresis in his affected hand.
* People with sensitivity alterations as a result of stroke.
* Evolution: subacute patients (from three months to one year, and who at the same time meet the subacute criteria of the IMSERSO document of the model of care for people with brain damage, as well as chronic patients (after one year, and who meet the chronicity criteria of the IMSERSO document of the model of care for people with brain damage).
* People without other concomitant pathologies that affect mobility and / or sensitivity
* The acceptance and signing of the informed consent by the user.
* Present a score equal to or greater than 24 points in the Mini-Mntal State Examination (MMSE).

  * Patients can be admitted or outpatient as long as they meet the above criteria and belong to the advanced neurorehabilitation unit.

Exclusion Criteria:

* Patients with Aphasia and / or Apraxia.
* Patients with serious difficulties in communication.
* Patients who do not present limitation of mobility and / or sensitivity.
* Other concomitant diseases.
* Diagnosis: left or posterior hemisphere stroke.
* Scores less than 24 points on the MMSE.
* Age over 80 years and under 30 years.
* The non-acceptance and signing of the informed consent by the subject.
* Evolution: acute patients less than three months of evolution.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-15 (Estimated); Primary Completion 2021-05-15 (Estimated); Study Completion 2021-06-15 (Estimated)

PRIMARY OUTCOMES:
Change from Fugl Meyer Assessment scale for the upper limb (change): Pre-treatment | Pre-treatment
  Motor Function
Change from Fugl Meyer Assessment scale for the upper limb at 1,5 months (change): Post-treatment period | Post-treatment (1,5 months)
  Motor Function

SECONDARY OUTCOMES:
Semmes-Weinstein ® monofilaments for sensitivity assessment | One month and a half
  Sensitivity. 0: no sensitivity. 1: alteration sensitivity. 2: normal. Higher scores mean a better outcome
Motor Activity Log | One month and a half
  Functionality. MAL scale is scored on six points, ranging from zero (never used) to five (the same as pre-stroke), and participants may select halfway scores, such as 1.5. Before its administration, the differences between the AOU and QOM scales were explained in detail and, during the test administration, these differences were emphasized at regular intervals. Higher scores mean a better outcome
Stroke Impacte Scale. | One month and a half
  Quality of life. The SIS version 3.0 includes 59 items and assesses 8 domains:
  Strength - 4 items Hand function - 5 items ADL/IADL - 10 items Mobility - 9 items Communication - 7 items Emotion - 9 items Memory and thinking - 7 items Participation/Role function - 8 items An extra question on stroke recovery asks that the client rate on a scale from 0 - 100 how much the client feels that he/she has recovered from his/her stroke. Higher scores mean a better outcome
Questionnaire of satisfaction with technology | One month and a half
  Satisfaction. Likert scale related to satisfaction. Total: 50 points. Higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. OMS. Who Steps Stroke Manual. En: Manual de la OMS para la vigilancia de accidentes cerebrovasculares. OMS 2006; p.1-5. 2. Pinedo S, De la Villa FM. Complicaciones en el paciente hemipléjico durante el primer año tras el ictus. Rev Neurol 2001; 32: 206-9. 3. Steultjens E, Dekker J, Bouter L, Van des Nes J, Van den Ende C, Landi F et al. Occupational Therapy for Stroke Patients: A systematic Review. Occupational Therapy for Stroke Patients: When, Where and How? Stroke 2003; 34; 676-87. 4. Brea A, Laclaustra M, Martorell E, Pedragosa À. Epidemiología de la enfermedad vascular cerebral en España. Clin e Investig en Arterioscler. 2013;25(5):211-7. 5. Cuadrado Á. Rehabilitación del ACV: evaluación, pronóstico y tratamiento Rehabilitation of the stroke: evaluation, prognosis and treatment. GaliciaclinicaInfo 2009;70(3):1-40. 6. Larsen LH, Zibrandtsen IC, Wienecke T, Kjaer TW, Christensen MS, Nielsen JB, et al. Corticomuscular coherence in the acute and subacute phase after stroke. Clin Neurophysiol 2017;128(11):2217-26. 7. Murphy MA, Resteghini C, Feys P, Lamers I. An overview of systematic reviews on upper extremity outcome measures after stroke. BMC Neurol. 2015 Mar 11;15(1). 8. Wu CY, Huang PC, Chen YT, Lin KC, Yang HW. Effects of mirror therapy on motor and sensory recovery in chronic stroke: a randomized controlled trial. Arch Phys Med Rehabil. 2013; 94:1023-30. 9. Invernizzi M, Negrini S, Carda S, Lanzotti L, Cisari C, Baricich A. The value of adding mirror therapy for upper limb motor recovery of subacute stroke patients: a randomized controlled trial. Eur J Phys Rehabil Med. 2013; 49:311-7. 10. Levin MF, Weiss PL, Keshner EA. Emergence of virtual reality as a tool for upper limb rehabilitation: incorporation of motor control and motor learning principles. Phys Ther. 2015; 95:415-25. 11. Sanchez Blanco. Monografico sobre Rehabilitacion de pacientes tras accidente cerebrovascular. Rehabilitacion (Madr). 2000; 36: 395-18. 19 12. Escuela Leeanne M. Carey de Ciencias de la Salud del Comportamiento, Universidad La Trobe, Victoria, Australia). 13. Sánchez-Blanco I, López de Munaín L, Ochoa-Sangrador C. Clasificación pronóstica de pacientes hemipléjicos: valor pronóstico en rehabilitación. Mapfre Med 1996; 7:187-96. 14. Sanchez Blanco. Predictive Model of functional independence in stroke patients admitted to a rehabilitation programme. Clin Rehabil. 1999; 13:464-75. 15. Subramanian S, Knaut LA, Beaudoin C, McFayden BJ, Feldman AG, Levin MF. Virtual reality environments for post-stroke arm rehabilitation. J Neuroeng Rehabil 2007; 4: 20. 16. Schmidth AR, Lee DT. Motor control and learning. A behavioural emphasis. Champaign. Human Kinetics; 1982. 17. Cano de la Cuerda R, Collado S. Neurorrehabilitacion. Métodos específicos de valoración y tratamiento. Madrid. Editorial Médica Panamericana; 2012: 89-139. 18. .Halsband U, Lange RK. Motor learning in man: a review of functional and clinical studies. J Physiol Paris. 2006; 99:414-24. 19. Langhorne P, Bernhardt J, Kwakkel G. Stroke rehabilitation. Lancet. 2011; 377:1693-702. 20. Park Y, Chang M, Kim KM, An DH. The effects of mirror therapy with tasks on upper extremity function and self-care in stroke patients. J Phys Ther Sci. 2015; 27:1499-501. 21. ZanYue et al. Hand Rehabilitation Robotics on Poststroke Motor Recovery. Behavioural Neurology Volume 2017. 22. Stein J, Bishop L, Gillen G, Helbok R. Robot-assisted exercise for hand weakness after stroke. A pilot study. American Journal of Physical Medicine & Rehabilitation. 2011; 90(11):887-894. 23. Celadon N, Dosen S, Binder I, Ariano P, Farina D. Proportional estimation of finger movements from high-density surface electromyography. Journal of Neuroengineering and Rehabilitation. 2016; 13(1):73. 24. Gandolfi M, Valè N et al. Effects of High-intensity Robot-assisted Hand Training on Upper Limb Recovery and Muscle Activity in Individuals With Multiple Sclerosis: A Randomized, Controlled, SingleBlinded Trial. Front. Neurol. 2018 Oct 24; 9:905. 25. Flor H. Cortical reorganisation and chronic pain: implications for rehabilitation. J Rehabil Med 2003; 41: 66-72. 26. Kishor L, Abigail W, Viswanathan R, John G. et al. Application of vibration to wrist and hand skin affects fingertip tactile sensation. Physiol Rep, 3 (7), 2015. 27. Collins DF, Refshauge KM, Todd G, Gandevia SC. Cutaneous receptors contribute to kinesthesia at the index finger, elbow, and knee. J Neurophysiol 2005; 94:1699-706. 11.